CLINICAL TRIAL: NCT07188584
Title: A Multicenter, Phase III Non-Inferiority Clinical Trial: Locoregional Volume-Reduction Versus Conventional Definitive Target IMRT Following Full-Dose Chemotherapy for Treatment-Naïve Distant Metastatic Nasopharyngeal Carcinoma Undergoing Full-Course Immunotherapy
Brief Title: Phase III Non-Inferiority Trial: Reduced-Target vs. Full-Target IMRT After Chemo in Immunotherapy-Treated Metastatic Nasopharyngeal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ming-Yuan Chen (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Cancer Hospital of Guangxi Medical University (Other); Fujian Cancer Hospital (Other Government); The Affiliated Cancer Hospital of Xiangya School of Medicine Central South University (Unknown); Sun Yat-sen University Cancer Center, Sun Yat-sen University (Unknown); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Zhejiang Cancer Hospital (Other); West China Hospital (Other); Xiangya Hospital of Central South University (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other); Yunnan Cancer Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Wuzhou Red Cross Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other); Southern Medical University, China (Other)
Responsible Party: Sponsor-Investigator, Ming-Yuan Chen, Professior, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY[2025] Lunzi No. (K66)
Record Dates: First submitted 2025-08-03; First posted 2025-09-23 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: Distant Metastasis Nasopharyngeal Carcinoma; Full Course Immunotherapy; Reduced-Target Radiotherapy; Full-dose Chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced-Target Radiotherapy after Full-dose Chemotherapy under Full-course Immunotherapy (Experimental): Immunotherapy: Patients received maintenance treatment with PD-1 monoclonal antibody (a 3-week course as one cycle) until disease progression or reach 2 years.
  Chemotherapy: Platinum-containing doublet chemotherapy (before enrollment, 4-6 cycles) and concurrent cisplatin during radiotherapy.
  Radiotherapy: Patients received intensity-modulated radiotherapy technology. Experimental group: GTVnx: 69.96 Gy/33 Fr/2.12 Gy; GTVnd: 69.96 Gy/33 Fr/2.12 Gy; CTV1: 60.60 Gy/33 Fr/1.82 Gy; GTV2: No prescription dose (only delineated, actual dose is scattered dose).
  Interventions: Radiation: Reduced-Target Radiotherapy
- Conventional Full-Target Radiotherapy after Full-dose Chemotherapy under Full-course Immunotherapy (Active Comparator): Immunotherapy: Patients received maintenance treatment with PD-1 monoclonal antibody (a 3-week course as one cycle) until disease progression or reach 2 years.
  Chemotherapy: Platinum-containing doublet chemotherapy (before enrollment, 4-6 cycles) and concurrent cisplatin during radiotherapy.
  Radiotherapy: Patients received intensity-modulated radiotherapy technology. Control group: GTVnx: 69.96 Gy/33 F/2.12 Gy; GTVnd: 69.96 Gy/33 F/2.12 Gy; CTV1: 59.4 Gy/33 F/1.8 Gy; CTV2: 54 Gy/33 F/1.64 Gy.
  Interventions: Radiation: Conventional Full-Target Radiotherapy

INTERVENTIONS:
Radiation: Reduced-Target Radiotherapy — Experimental group: GTVnx: 69.96 Gy/33 Fr/2.12 Gy; GTVnd: 69.96 Gy/33 Fr/2.12 Gy; CTV1: 60.60 Gy/33 Fr/1.82 Gy; GTV2: No prescription dose (only delineated, actual dose is scattered dose).
  Arms: Reduced-Target Radiotherapy after Full-dose Chemotherapy under Full-course Immunotherapy
Radiation: Conventional Full-Target Radiotherapy — Control group: GTVnx: 69.96 Gy/33 F/2.12 Gy; GTVnd: 69.96 Gy/33 F/2.12 Gy; CTV1: 59.4 Gy/33 F/1.8 Gy; CTV2: 54 Gy/33 F/1.64 Gy.
  Arms: Conventional Full-Target Radiotherapy after Full-dose Chemotherapy under Full-course Immunotherapy

SUMMARY:
In order to further verify the effectiveness of the new prevention irradiation model for low-risk areas for nasopharyngeal carcinoma under immunotherapy, our team intends to conduct a non-inferiority clinical trial. The aim is to evaluate the efficacy and safety of two treatment modalities - local region reduced-target radiotherapy versus full-target radiatiotherapy (with/without CTV2) for newly diagnosed distant metastasis nasopharyngeal carcinoma, based on the full-course immunotherapy and full-dose chemotherapy. The primary endpoints are 2-year PFS and the incidence of grade 3 or higher radiation-related adverse events. If non-inferiority is confirmed, a new standard of "immunotherapy combined with reduced-target radiotherapy" will be established, ensuring efficacy while significantly reducing toxicity, and providing a more optimal comprehensive treatment strategy for nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma is a highly prevalent malignant tumor in the southern regions of China, with approximately 4% to 10% of patients presenting with distant metastasis at the initial diagnosis. The five-year survival rate of traditional sole systemic chemotherapy is less than 10%, and there is an urgent need to explore more effective treatment strategies. Our team previously conducted a single-center study (402 cases) and a national multicenter retrospective study (794 cases) and first revealed that local regional radiotherapy combined with systemic chemotherapy resulted in a 60% reduction in mortality compared to systemic chemotherapy alone (HR = 0.40) (Chen MY, Chin J Cancer, 2013; Eur J Cancer, 2015). To verify this finding, with the support of the 5010 project of Sun Yat-sen University, our team initiated the world's first phase III prospective clinical trial for newly diagnosed distant metastatic nasopharyngeal carcinoma in 2014. This trial confirmed that after 6 courses of adequate systemic chemotherapy, the control group was followed up, while the experimental group received local regional full-target area adequate radiotherapy, covering the gross tumor volume (GTV), high-risk clinical target area 1 (CTV1), and low-risk clinical target area 2 (CTV2), with a total radical dose of 70 Gy, 60 Gy and 54 Gy for prophylactic radiotherapy, extending the median progression-free survival (mPFS) from 6.7 months to 12.4 months, and the 2-year PFS rate from 3.6% to 35.0%. This "adequate chemotherapy + full-target adequate radiotherapy" dual-model achieved the "Global ASCO 17 Major Clinical Oncology Breakthrough" by the American Society of Clinical Oncology in 2021, directly promoting the inclusion of local radiotherapy in the standard recommended treatment for metastatic nasopharyngeal carcinoma in the US NCCN treatment guidelines, European ESMO guidelines, Chinese CSCO guidelines and CACA guidelines (Chen MY, JAMA Oncology, 2020).

With the widespread application of PD-1 monoclonal antibodies, GP chemotherapy combined with immunotherapy (with a maximum mPFS of 21.4 months and 2-year PFS of 44.8%) has become the first-line chemotherapy regimen for recurrent/metastatic nasopharyngeal carcinoma. However, these single-drug studies did not combine local-region radiotherapy, and its value in newly diagnosed distant metastatic nasopharyngeal carcinoma has not been optimized. Therefore, our team further conducted a phase II clinical trial, sequentially administering local-region full-target radiotherapy and PD-1 monoclonal antibody during and after systemic adequate chemotherapy, and the results showed that the mPFS exceeded 30.6 months, and the 2-year PFS rate reached 54%, confirming the outstanding efficacy of the "adequate chemotherapy + half-course immunotherapy + full-target radiotherapy" triple model (Chen MY, Cell Reports Medicine, 2023).

However, the preventive irradiation area CTV2 in full-target radiotherapy has a wide coverage and is irradiated with a dose of 54 Gy or more, resulting in a 33.9% incidence of grade 3 acute mucositis and 5.2% of late hearing damage and other adverse events, severely restricting treatment tolerance. Moreover, basic research has revealed that lymph node integrity is crucial for immunotherapy, and excessive destruction of draining lymph nodes (>30 Gy) will deplete the Tim-3-TCF-1⁺ CD8+ T cell subset (with stem cell characteristics, driving long-term responses to PD-1 monoclonal antibodies), while weakening the ability of antigen-presenting cells to activate T cells, leading to impaired systemic anti-tumor immunity. Clinical retrospective analysis also indicates that patients undergoing extensive preventive lymph node dissection who received PD-1 monoclonal antibody treatment had significantly shorter PFS (HR = 0.46). Based on this, we propose the following hypothesis: In the era of immunotherapy, omitting the traditional CTV2 for the irradiation area, and exempting the low-risk invasion area of the primary lesion and the lymphatic drainage areas such as the neck II-IV zone from the preventive irradiation, can not only reduce toxicity but also preserve the lymph node immune microenvironment, thereby potentially enhancing the systemic anti-tumor response and being more conducive to the control of systemic metastatic lesions. Therefore, our team has further carried out a phase II clinical trial. After 6 courses of full-dose chemotherapy and immunotherapy, sequential local-region reduced-CTV2 radiotherapy and concurrent and maintenance immunotherapy of PD-1 monoclonal antibody were administered. The results showed that the 1-year PFS rate was as high as 77%, preliminarily suggesting that the "full-dose chemotherapy + full-course immunotherapy + reduced target radiotherapy" new triad model may be superior to the conventional full-target radiotherapy original triad model.

To further verify the effectiveness of this new model, our team intends to conduct the world's first phase III non-inferiority clinical trial for the initial treatment of advanced nasopharyngeal carcinoma. Patients with newly diagnosis distant metastatic nasopharyngeal carcinoma who respond sensitively to chemoradiotherapy will be included. Under the full-course PD-1 treatment, they will randomly receive reduced-target radiotherapy (GTV + CTV1) or full-target radiotherapy (GTV + CTV1 + CTV2). The primary endpoints are the 2-year PFS rate (non-inferiority threshold HR = 1.5) and the incidence of grade 3 or higher radiotherapy-related adverse events.

The innovation of this research lies in: pioneering a new radiotherapy strategy under nasopharyngeal carcinoma immunotherapy that exempts the preventive irradiation of low-risk areas; revealing the mechanism correlation between reduced-target radiotherapy and the dynamics of immune cell subgroups; providing evidence-based evidence for "minimal irradiation" in immunotherapy for solid tumors.

If the study confirms non-inferiority, it will achieve three major translational values: clinical level, establishing a new standard of "reduced-target radiotherapy - immune synergy"; scientific level, clarifying the regulatory role of lymph node microenvironment in radiotherapy and immunotherapy; social level, optimizing the allocation of medical resources by improving the quality of life of patients and their treatment compliance. The implementation of this study will challenge the traditional full-target radiotherapy paradigm, providing a more efficient and less toxic reduced-target radiotherapy scheme for metastasis nasopharyngeal carcinoma, as well as locally advanced nasopharyngeal carcinoma and even other solid tumors, with significant clinical and scientific significance.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years - 70 years.
* The patient has signed the informed consent form and is willing and able to follow the visit schedule, treatment plan, laboratory tests and other research procedures as per the research plan.
* Newly diagnosed distant metastasis patients who achieved complete response (CR) or partial response (PR) after receiving adequate first-line systematic therapy (platinum-containing doublet chemotherapy + PD-1 monoclonal antibody).
* Nasopharyngeal carcinoma non-keratinizing carcinoma (differentiated or undifferentiated type, i.e., WHO type II or III), confirmed by histological and/or cytological examination, with metastatic lesions detected on imaging (biopsy of metastatic tissue is preferred but not mandatory).
* Clinical stage: TanyNanyM1, stage IVB (AJCC 9th edition).
* ECOG score: 0-1.
* Female subjects with reproductive capacity must have a negative urine or serum pregnancy test within 7 days prior to enrollment, and must agree to take effective contraceptive measures during the study.
* For male subjects, if the female partner still has reproductive capacity, the male subject must agree to take effective contraceptive measures during the study.

Exclusion Criteria:

* Patients with malignant pleural effusion or those with other malignant tumors
* Patients who have received ≥2 prior lines of systemic therapy.
* Patients with known or suspected autoimmune diseases, including dementia and epileptic seizures.
* Patients with grade ≥ II coronary heart disease, arrhythmia (including QTc interval prolongation in males > 450 ms, females > 470 ms) and heart failure.
* Patients who received systemic or local glucocorticoid treatment within 4 weeks prior to enrollment.
* Patients with comorbidities requiring long-term use of immunosuppressive drugs or requiring systemic or local use of corticosteroids at immunosuppressive doses.
* Patients with active pulmonary tuberculosis (TB), who are undergoing anti-TB treatment or have received anti-TB treatment within 1 year prior to screening.
* HIV-positive individuals; HBsAg positive and HBV DNA copy number positive (quantitative detection ≥ 1000 cps/ml); chronic hepatitis C blood screening positive (HCV antibody positive).
* Patients who received any anti-infective vaccine (such as influenza vaccine, varicella vaccine, etc.) within 4 weeks prior to enrollment.
* At the time of randomization, the expected lifespan of the patients was less than 6 months.
* Other patients deemed unsuitable for inclusion by the treating physicians.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
2-year Progression-Free Survival (PFS) | 2 years
  The PFS was defined as the duration from the date of random assignment to the date of disease progression or censored at the date of the last follow-up.
The incidence rate of radiotherapy-related ≥ grade 3 adverse events | 2 years
  Including the evaluation of acute subjective and objective toxic reactions as well as the evaluation of late subjective toxic reactions. The NCI-CTC 5.0 standard and RTOG standard were adopted.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | 2 years
  Defined as the proportion of patients who, after receiving treatment, have achieved complete response (CR) or partial response (PR) and maintain this state for a certain period of time (evaluated by the investigator according to RECIST 1.1)
Disease control rate (DCR) | 2 years
  Defined as the proportion of patients who achieve CR + PR + SD after receiving treatment, and maintain this state for at least 4 weeks.
Overall survival time (OS) | 2 years
  Defined as the time interval from the start of randomization, due to any cause, death occurs (if no death, censored at the last known survival date).
Health-related Quality of Life | 2 years
  Changes from baseline in patient-reported quality of life scores assessed every 2 cycles using the EORTC QLQ-C30 questionnaire (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, version C30). The scores range from 0 to 100, with higher scores indicating a better quality of life outcome.
Adverse Events Reporting | 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Head and Neck Cancer-Specific Quality of Life | 2 years
  Changes from baseline in head and neck cancer-specific symptoms and functions assessed every 2 cycles using the EORTC QLQ-H&N35 module (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Head and Neck Cancer Module). The scores range from 0 to 100, with higher scores indicating a better quality of life outcome and lower scores indicating worse symptoms or functions.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong 519000 Recruiting, Zhuhai, China